CLINICAL TRIAL: NCT02145702
Title: Impact of Exercise on Cognitive Impairment in End-Stage Renal Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding has expired
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Aditi Gupta, MD, Assistant Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000284
Record Dates: First submitted 2014-05-17; First posted 2014-05-23 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Cognitive Impairment; End-Stage Renal Disease
Keywords: ESRD; Kidney Failure; Exercise; Cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Kidney Failure, Chronic; Renal Insufficiency; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Group (Experimental): Subjects randomized to this group will start 12 weeks of supervised aerobic exercise after baseline testing.
  Interventions: Other: Aerobic Exercise
- Control Group (Experimental): Subjects randomized to this group will continue with 12 weeks of Standard Care. After 12 weeks, the subjects will cross over to the exercise arm and undergo baseline testing again and then start 12 weeks of exercise intervention.
  Interventions: Other: Aerobic Exercise; Procedure: Standard Care Dialysis

INTERVENTIONS:
Other: Aerobic Exercise — Each exercise session will be conducted at the KUMC Exercise and Cardiovascular Health (REACH) Laboratory. Exercise sessions will include a warm-up period, exercise period and a cool down period. Exercise intervention individualized based on health of participant. Subject will be asked to completed two exercise sessions per week for 12 weeks.
Procedure: Standard Care Dialysis — 12 weeks of standard of care.
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the impact of 12 weeks of exercise on cognition in patients with end stage renal disease.

DETAILED DESCRIPTION:
Patients with end stage renal disease have higher cognitive impairment than general population. They also have decreased physical and functional capacity. Exercise has shown to improve cognition in general population. This study will evaluate if exercise improves cognition in dialysis patients. It will also evaluate whether exercise affects performance in daily activities, mood or depression and inflammatory markers in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESRD on dialysis
* Age greater than 20 years
* Have means of transportation to and from the exercise session
* Speak English (as the neuropsychological tests will be performed in English)

Exclusion Criteria:

* Recent myocardial infarction (within 6 weeks), unstable angina, uncontrolled arrhythmias, congestive heart failure (> NYHA grade II)
* History of stroke in the last 2 months
* Active respiratory disease
* Uncontrolled hypertension
* Severe uncontrolled diabetes
* Persistent predialysis hyperkalemia
* Active decompensated liver disease
* Symptomatic peripheral vascular disease
* Musculoskeletal abnormalities that will be prohibit their participation in the exercise program
* Health conditions needing frequent hospitalizations
* Other health conditions causing inability to follow exercise program correctly
* Unwillingness to participate in structured exercise program
* Current use of antipsychotics or anti-epileptics
* Inability to hear, read or write which will limit their ability to perform the cognitive tests

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Feasibility | Up to 26 Weeks
  Subject compliance with exercise training

SECONDARY OUTCOMES:
Cognitive function | Baseline, within1 week before and within 1 week after exercise intervention
  Measured using a standard battery of neuropsychological tests.
Markers of inflammation | Baseline, within 1 week before and within 1 week after exercise intervention
  Markers of inflammation will be evaluated before and after exercise intervention

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Gupta, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States